CLINICAL TRIAL: NCT02942732
Title: Effect of Treating Vitamin D Deficiency on Glucose Homeostasis and Metabolic Markers in Apparently Healthy, Young or Aged, Normal-weight or Obese Lebanese People
Brief Title: Vitamin D Supplementation and Glycemic Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université d'Auvergne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UAuvergne
Record Dates: First submitted 2016-10-16; First posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Insulin Resistance
Keywords: Vitamin D; Glucose; HbA1C; Insulin resistance; Blood lipids
MeSH Terms: conditions — Insulin Resistance | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- normal-weight adult subjects (Other): normal-weight adult subjects (n=30, age ≤ 65 years and BMI ≤ 25 kg/m²) All assigned patients received a supplement of 10,000 IU cholecalciferol (Euro-Pharm International, Canada) to be taken three times per week. The treatment was led for a period of 6 months.
  Interventions: Dietary Supplement: cholecalciferol (Euro-Pharm International, Canada)
- overweight adult subjects (Other): overweight adult subjects (n=30, age ≤ 65 years and BMI ≥ 25 kg/m²) All assigned patients received a supplement of 10,000 IU cholecalciferol (Euro-Pharm International, Canada) to be taken three times per week. The treatment was led for a period of 6 months.
  Interventions: Dietary Supplement: cholecalciferol (Euro-Pharm International, Canada)
- normal-weight elderly (Other): normal-weight elderly (n=60, age ≥ 65 years and BMI ≤ 25 kg/m²) All assigned patients received a supplement of 10,000 IU cholecalciferol (Euro-Pharm International, Canada) to be taken three times per week. The treatment was led for a period of 6 months.
  Interventions: Dietary Supplement: cholecalciferol (Euro-Pharm International, Canada)
- overweight elderly (Other): overweight elderly (n=60, age ≥ 65 years and BMI ≥ 25 kg/m²) All assigned patients received a supplement of 10,000 IU cholecalciferol (Euro-Pharm International, Canada) to be taken three times per week. The treatment was led for a period of 6 months.
  Interventions: Dietary Supplement: cholecalciferol (Euro-Pharm International, Canada)

INTERVENTIONS:
Dietary Supplement: cholecalciferol (Euro-Pharm International, Canada) — All assigned patients received a supplement of 10,000 IU cholecalciferol (Euro-Pharm International, Canada) to be taken three times per week. The treatment was led for a period of 6 months.

SUMMARY:
The investigators examined the effect of vitamin D supplementation on glucose homeostasis and metabolic markers in healthy normal weight and overweight young subjects and healthy normal-weight and overweight elderly subjects living in Beirut, Lebanon.

DETAILED DESCRIPTION:
A low serum 25-hydroxyvitamin D (25(OH)D) concentration has been shown to correlate with higher fasting blood glucose (FBG) and insulin levels and other metabolic abnormalities like dyslipidemia. Previous studies suggest that vitamin D supplementation is able to improve insulin sensitivity and metabolic markers. The aim of the study was to investigate the effect of vitamin D supplementation on glucose homeostasis and metabolic markers in healthy normal weight and overweight young subjects and healthy normal-weight and overweight elderly subjects living in Beirut, Lebanon. Participants (n= 180; 93 men and 87 women) deficient in vitamin D were recruited from Saint Charles Hospital, Beirut, Lebanon. Four groups were recruited: normal-weight adults (n=30, age ≤ 65 years and BMI < 25 kg/m²), overweight adults (n=30, age ≤ 65 years and BMI ≥ 25 kg/m²), normal-weight elderly (n=60, age ≥ 65 years and BMI < 25 kg/m²) and overweight elderly (n=60, age ≥ 65 years and BMI ≥ 25 kg/m²).

Participants received a supplement of 10,000 IU cholecalciferol to be taken three times per week for a period of 6 months. Glucose homeostasis and metabolic markers were measured at start of treatment, at 3 months and at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants with no medical history of congestive heart failure, acute heart insufficiency and renal failure were included

Exclusion Criteria:

* Participants with medical history of congestive heart failure, acute heart insufficiency and renal failure were excluded

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2013-02; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Fasting blood glucose (mmol/l) | Baseline and 6 months
  Change in Fasting blood glucose in mmol/l
HbA1C (%) | Baseline and 6 months
  Change in HbA1C (%)
HOMA-IR | Baseline and 6 months
  Change in HOMA-IR
Fasting Insulin (mIU/L) | Baseline and 6 months
  Change in Fasting Insulin (mIU/L)

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Walrand, PhD, Study Director — Auvergne Univeristy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Nagpal J, Pande JN, Bhartia A. A double-blind, randomized, placebo-controlled trial of the short-term effect of vitamin D3 supplementation on insulin sensitivity in apparently healthy, middle-aged, centrally obese men. Diabet Med. 2009 Jan;26(1):19-27. doi: 10.1111/j.1464-5491.2008.02636.x. PMID 19125756
- [Result] Pittas AG, Lau J, Hu FB, Dawson-Hughes B. The role of vitamin D and calcium in type 2 diabetes. A systematic review and meta-analysis. J Clin Endocrinol Metab. 2007 Jun;92(6):2017-29. doi: 10.1210/jc.2007-0298. Epub 2007 Mar 27. PMID 17389701